CLINICAL TRIAL: NCT03636672
Title: The Effects of Bicycle Simulator Training on Anticipatory and Compensatory Postural Control in Older Adults: A Randomized Controlled Trial
Brief Title: Bicycle Simulator Training in Older Adults: A Randomized Controlled Trial
Acronym: PerStBiRo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BARZI0104
Record Dates: First submitted 2018-07-22; First posted 2018-08-17 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Accidental Falls
Keywords: falls; Balance control; Aging; Balance reactions; Perturbation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Perturbation training during stationary bicycle riding
  Interventions: Procedure: perturbation training
- control (Active Comparator): stationary bicycle riding training
  Interventions: Procedure: perturbation training

INTERVENTIONS:
Procedure: perturbation training — perturbation training during stationary bicycle riding

SUMMARY:
A Randomized Control Trial will be conducted with Independent old adults (age 70 years old and older) who willing to participate in the study. They will be randomly allocated to two groups: 1) Stationary bicycle riding that includes perturbation balance training during riding; 2) Stationary bicycle riding that does not includes perturbation balance training during riding. Balance and Gait assessments will be tested before and after 3 months of training (2-3 times a week).

DETAILED DESCRIPTION:
Falls and fall-related injuries are common elder health problems. Falls are the leading cause of fatal and nonfatal injuries among older adults, reducing mobility and independence, and increase the risk of death. Between 30 to 40% of the community-dwelling older persons fall at least once a year, usually by falling sideways that is resulting in 95% of hip fractures. In the U.S. in 2014, the estimated direct medical costs for fall-related injuries were $31.3 billion and is expected to reach $67.7 billion by 2030 Age-related changes in the balance control system increase the risk of falls. Execute a rapid step, whether voluntary or compensatory, is the most important balance strategy to prevent a fall. In voluntary stepping test, the foot contact times (i.e., stepping time) and reaction time (initiation phase) were able to predict future fall and injury from fall. Studies of the reactive postural control have shown that older adults initiate stepping at lower levels of instability, use multiple steps, experience leg collisions or fail to recover balance compared to younger adults. The Medio-Lateral center of pressure sway range with Eyes Closed is the best single predictor for future fall.

Studies showed that older adults were able to adapt in a reactive manner after participation in a Perturbations based balance training (PBBT) that challenged the mechanisms responsible for dynamic stability. These studies also showed a reducing in rate of falls and diverse risks of falls in older adults (voluntary stepping times, balance control in standing and walking, improved function and reduced fear of falls). however, in these studies the training devices and programs were designed to participants who able to walk independently the whole training sessions, lasting 20-45 minutes each and appropriate only for a small portion of the general elderly population. In fact, in 2014 in U.S., the community-dwelling older persons that reported a fall were divided equally into three health status: poor-fair, good, very good-excellent with 33% rate of fall each subgroup. This fact motivates us to provide accessibility PBBT for a wider range of the elderly population, and not for the "strongest" older subjects.

Inspired by the well-known health advantages of cycling and the medio-lateral postural control demand during two-wheel bicycle riding, encourage us to conduct a preliminary study for feasibility. In this study we found older adults who aged with bicycle riding habits have benefits in reactive and predictive aspects of postural control mechanisms (particularly in the medio-lateral postural control) while standing and stepping, both related to risk of falling in the elderly (see Preliminary result section). Because the special importance of the medio-lateral balance control for preventing lateral falls and hip fractures in old age, considering our preliminary findings, we hypothesize that following exposure to training program that includes unexpected perturbations exercises during cycling will significantly improve compensatory and voluntary stepping times as well as the medio-lateral balance control in older adults, factors that are associated with falls and fall- related injuries.

Objectives: firstly, to explore whether training while riding a new bicycle simulator device providing unexpected perturbations can reduce risks of falls in standing and walking in independent older adults. Secondly, if so, to examine this bicycle simulator device providing unexpected perturbations method in a wider range of elderly subjects (i.e., who do not walk independently or walk for only short distances or with assisted devices or suffering from fear of falling or in pre-walking rehabilitative phases after stroke or other morbidity).

Methods Study design: A double blinded randomized controlled trial. Participants: Relatively healthy Community dwelling older adults that are 70 years or older, independent in daily living activities, walking without assistive devices, without morbidity that influence balance performance. The study will be approved by the Helsinki committee of Barzilai University medical center, Ashkelon, Israel. All subjects will sign an informed consent statement.

Training programs: We will use two identical exercise bicycles, one will remain a stationary Bicycle device for the control group, and bicycle simulator device providing unexpected perturbations during a bicycle simulator riding for the experimental group. The intervention Group will receive 24 bicycle simulator device providing unexpected perturbations sessions, twice a week for 12 weeks (about 20 min. each). The subjects will be instructed to "ride on the bicycle in your preferred pace and try to stabilize yourself". To prevent injury if loss of balance occurred during the cycling, the subject will wear a loose safety harness that can arrest the fall. The bicycle simulator device providing unexpected perturbations program will have 24 levels of difficulty with increasing levels of perturbations (i.e., increase displacement, velocity and accelerations of the translations). The control group will receive 24 sessions, twice a week for 12 weeks, about 20 minutes' bicycle riding on the stationary device, pedaling in subject own preferred pace without perturbations and wearing a loose safety harnesses. Since both group will train on two identical exercise bicycles, they will be blinded to the allocation to intervention or control group.

Assessments: 1) Compensatory Step Execution tests during Standing and Walking: The subjects will be instructed to react naturally. Ten perturbation levels will be induced through a device that provides controlled and unexpected anterior-posterior and medio-lateral platform translations during a single belt treadmill in standing and walking. Four directional perturbations (right/left/forward/backward) in a random order each level for a total of 40 perturbation trials. Kinematic analysis: Three-dimensional kinematic data will be collected through the optical motion capture, providing kinematic analysis of a motion sequence. Sixteen infrared cameras are covered the lab space sample simultaneously, at frequency of 200 Hz, the location of 35 reflective markers placed on anatomical landmarks of the body and another two on the moving platform. The following Balance compensatory kinematics parameters: (1) Platform perturbation; (2) First Step initiation time (milliseconds); (3) Foot contact time (milliseconds); (4) Compensatory Step execution time (milliseconds); (5) Step swing time (milliseconds); (6) Step length (centimeters); (7) End of Compensatory steps time (milliseconds); (8) Total distance center of mass made (centimeters); (9) Distance of center of mass from leg at the step-beginning point (centimeters); 10) Arms lift initiation times (milliseconds); 11) Maximal arms swing amplitude/length (centimeters); 12) Arms swing times (milliseconds). Observational analysis: observing each trail video and identifying the compensatory reactions (see preliminary results). 2) Voluntary Step Execution Test: Participants are instructed to voluntary step as quickly as possible following a somatosensory cue, given randomly on one of their feet. A total of 8 trials will be conducted in singe task and dual task conditions (while performing the modified Stroop task). Specific temporal events were extracted from the step execution data: (a) Reaction Time; (b) Foot Contact Time; (c) Preparation Time; (d) Swing Time. 3) Postural Stability: The subjects will be instructed to stand barefoot as still as possible on the force platform in a standardized stance. Five 30-s quiet-standing trials with eyes open and five trails with eyes blindfolded. Evaluation of balance control will be made using both, traditional measure of postural sway (e.g. medio-lateral-sway, anterior-posterior -sway, sway velocity, and sway area), and calculating the Stabilogram-Diffusion Analysis parameters from center of pressure data. In addition, clinical measurements and questionnaires will be conducted as the secondary outcome measures: Berg Balance Scale (BBS); 6-minute walk test (6MWT); Medical History form; Late Life Function and Disability Instrument (LLFDI); Falls Efficacy Scale-International (FES); Mini Mental state examination (MMSE).

ELIGIBILITY:
Inclusion Criteria:

* age 70 and over
* able to walk independently
* The provision of a medical certificate from the family physician allowing participation in physical training that requires walking two or three times a week.

Exclusion Criteria:

* suffers from ischemic heart disease which will restrict exercise and chronic obstructive pulmonary disease and uncontrolled blood pressure;
* severe vision problems (blindness);
* mini-mental score of 24 or more;
* At least one year after hip or knee replacement surgery or after fractures of the lower extremities;
* Amputation on the lower limb.
* neurological diseases or after a stroke

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Compensatory Step Execution tests during Standing and Walking | change from baseline to 3 months later
  the time from perturbation to foot contact the floor completing the recovery stepping will be measured in milliseconds

SECONDARY OUTCOMES:
Postural Sway measure using force plate | change from baseline to 3 months later
  body sway will be measured to evaluate control of posture
Berg Balance Scale | change from baseline to 3 months later
  The berg balance score 14 performance based measures/subscales that are score from 0-4 of balance skills (the total score ranges is 0-56), higher score represent better balance.
6-minute walk test (6MWT); | change from baseline to 3 months later
  time of walking six minutes
Late Life Function and Disability Instrument (LLFDI); | change from baseline to 3 months later
  32 questions about how much dificult to perform a daily activities
Falls Efficacy Scale-International | change from baseline to 3 months later
  The fall efficacy scale measure includes 10 questions that evaluate the fear of fall during a daily activities (score ranged from 10-100). Higher values represent more fear of falling
Voluntary Step Execution Test | change from baseline to 3 months later
  voluntary stepping will be measured in milliseconds

CONTACTS AND LOCATIONS:
Locations (1):
- Ben-Gurion University of the Negev, Beersheba, Israel

REFERENCES:
- [Derived] Batcir S, Livne K, Lehman RL, Berdichevsky Y, Maoz S, Shkedy LW, Adar R, Rabaev E, Bachner YG, Shani G, Lubovsky O, Shapiro A, Alexander NB, Melzer I. Feedback-based perturbation balance training during stationary cycling improves reactive and proactive balance among older adults: a single-blinded randomised controlled trial. Age Ageing. 2025 Aug 1;54(8):afaf215. doi: 10.1093/ageing/afaf215. PMID 40794910
- [Derived] Batcir S, Lubovsky O, Bachner YG, Melzer I. The Effects of Bicycle Simulator Training on Anticipatory and Compensatory Postural Control in Older Adults: Study Protocol for a Single-Blind Randomized Controlled Trial. Front Neurol. 2021 Jan 18;11:614664. doi: 10.3389/fneur.2020.614664. eCollection 2020. PMID 33536998